CLINICAL TRIAL: NCT02231502
Title: Optimising Vegetable Based Convenience Food Production to Retain Compounds Found in Vegetables
Brief Title: Innovation in Food Production Techniques to Improve Bioactive Content
Acronym: ENRICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other); PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14/EE/0070
Record Dates: First submitted 2014-08-27; First posted 2014-09-04 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Bioavailability
Keywords: Bioavailability in healthy individuals

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Vegetable-based convenience food (Experimental): One time ingestion of a vegetable-based convenience product. Dietary restrictions will be observed (i.e. avoidance of some vegetables) for 3 days prior to the bioavailability assessment (a list of foods to avoid will be provided).
  At least 7 days wash-out between each assessment visit.
  Interventions: Other: Vegetable-based convenience food
- Vegetable meal (Active Comparator): One time ingestion of a minimally processed vegetable meal. Dietary restrictions will be observed (i.e. avoidance of some vegetables) for 3 days prior to the bioavailability assessment (a list of foods to avoid will be provided).
  At least 7 days wash-out between each assessment visit.
  Interventions: Other: Vegetable meal

INTERVENTIONS:
Other: Vegetable-based convenience food
  Arms: Vegetable-based convenience food
Other: Vegetable meal
  Arms: Vegetable meal

SUMMARY:
The purpose of this study is to establish to what extent innovations in food production techniques may facilitate retention of bioactive compounds in healthy individuals.

The study has a single-blinded (outcome assessor), cross-over design; wherein, the plasma concentration and urinary excretion levels of a range of bioactive compounds will be assessed over a 24 hour period following intake of either a vegetable based convenience food, or a minimally processed meal containing the same vegetable materials.

To do this, 20 healthy volunteers will attend two assessment days (and a follow-up assessment at +24hr) and will provide blood and urine samples, which will be collected at biologically relevant times over the 24 hour period. In this cross-over study, each meal will be eaten on separate days, with a wash-out period of at least 1 week between assessments.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* ≥ 18 years old
* Successful biochemical, haematological and urinalysis assessment at screening

Exclusion Criteria:

* Current smokers, or ex-smokers ceasing < 3 months ago
* Pregnant women, or those currently breast feeding
* Subjects with existing or significant past medical history of medical conditions likely to affect the study measures i.e. diabetes, hepatic, renal, digestive or cancer (excluding Basal-cell carcinoma) - to be judged by the study clinical advisor.
* Those unprepared to adhere to dietary restrictions for 3d preceding and during each assessment day.
* Parallel participation in another research project involving dietary intervention and/or sampling of biological fluids/material.
* Those on therapeutic diets or having experienced substantial weight loss (to be judged by clinical advisor) within 3 month of screening
* Taking dietary supplements containing flavonoids, isothiocyanates or carotenes (including multivitamins) (and unwilling to cease intake during, and 1 month preceding the trial) or unwilling to maintain existing intake of other supplements.
* Prescribed medications likely to affect ADME (absorption, distribution, metabolism, and excretion); medications to be assessed for suitability by the clinical advisor.
* Clinical advisor judged: abnormal biochemical, haematological or urinary results or measurements considered to be counter indicative for the study: including kidney and liver function, fasting glucose (especially if indicative of diabetes), lipid abnormalities, full blood count.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
24hr excretion of bioactive compounds | 24h
  A range of bioactive compounds found in vegetables, and their metabolites, will be assessed in blood and/or urine samples collected over a 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Aedin Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Norwich Medical School, Norwich, Norfolk, United Kingdom